CLINICAL TRIAL: NCT01665586
Title: Effective Dose of Dexmedetomidine for Sedation in Patients Undergoing TURP/TURB Under Spinal Anesthesia With or Without Fentanyl by Age Groups: Randomized Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2011-0927
Record Dates: First submitted 2012-07-31; First posted 2012-08-15 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Benign Prostate Hyperplasia; Bladder Tumor
Keywords: dexmedetomidine; sedation in elderly patient; spinal anesthesia
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Placebo Comparator): : Spinal anesthesia with 6mg bupivacaine and intrathecal placebo(normal saline) added
  Interventions: Drug: dexmedetomidine
- Group F (Active Comparator): : Spinal anesthesia with 6mg bupivacaine and intrathecal small dose of fentanyl(20micro gram)
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — Spinal anesthesia regimen Group F: 6mg bupivacaine + 20mcg fentanyl (intrathecal) + o.4 cc 5% dextrose water Group C: 6mg bupivacaine + 0.4 cc normal saline + 0.4cc 5% dextrose water
  dexmedetomidine 0.2~0.8 micro gram/kg intravenous administration after the sterilization of the spinal anesthesia level, and prehydration

SUMMARY:
Recently many studies reported that intraoperative dexmedetomidine administration undergoing spinal anesthesia give a satisfactory sedation in elderly patients and cause less respiratory depressions compared other sedatives(e.g. benzodiazepine) But the optimal dose of dexmedetomidine for sedative effect in elderly patients undergoing spinal anesthesia was not got general consensus.

The investigators hypothesized that the dose requirements would be lower than in elderly patients than young patients. Furthermore, intrathecal small dose opioids enhance the analgesia provided by bupivacaine due to synergistic effects and it would reduce the dose of dexmedetomidine.

The purpose of this study was to determine the dose of dexmedetomidine to provide satisfactory sedation undergoing spinal anesthesia with or without additive small dose intrathecal opioids.

Elderly patients(65~85 years old) undergoing TURP or TURB were enrolled in this single-blinded study. Forty patients were randomly assigned to receive intrathecal hyperbaric bupivacaine 6mg coadministered with 20mcg fentanyl or placebo normal saline 0.4cc. After the induction (bilateral T10 sensory level to pinprick within 5 mins of intrathecal drug administration), continuous intravenous dexmedetomidine was started in dose of 0.8, 0.6, 0.5, 0.4, 0.3, or 0.2mcg. Successful sedation was defined as OASS score 3 or 4 within 20 minutes of dexmedetomidine infusion. The dose of dexmedetomidine was selected for each patient according to an up and down method. Intraoperative arterial pressure, heart rate, and bispectral index was compared. Postoperative pain score, the time for the regression of sensory and motor was recorded for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65~85 years olds undergoing TURB or TURP.
* No contraindication of spinal anesthesia.
* ASA class I and II.
* Patients consented to spinal anesthesia were enrolled.

Exclusion Criteria:

* Patients with hypovolemia, coagulation disorders, local infection at the site of operation, history of headache, heart diseases, and history of allergy, chronic alcohol use or abuse, anemia, congenital heart diseases, bundle block, congestive heart failure or arrythmias, and patients who had recently received sedative drugs or were under antidepressant treatment were not included in the study.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Observer's Assessment of Alertness/Sedation scale, OAA/S | from 5 min after study drug (dexmedetomidine or placebo) adminstration to the ending point of surgery.
  Observer's Assessment of Alertness/Sedation scale, OAA/S 5 Responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly and/or repeatedly 2 Responds only after mild prodding or shaking
  1 Responds only after painful trapezius squeeze 0 No response after painful trapezius squeeze 0 No response after painful trapezius squeeze

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, and Anesthesia and Pain Research Institute, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Kim WO, Kim HB, Kil HK. Adequate sedation with single-dose dexmedetomidine in patients undergoing transurethral resection of the prostate with spinal anaesthesia: a dose-response study by age group. BMC Anesthesiol. 2015 Jan 27;15:17. doi: 10.1186/1471-2253-15-17. PMID 25971886